CLINICAL TRIAL: NCT06756399
Title: Relationship Between Sarcopenia and Peripheral and Respiratory Muscle Strength in Geriatric Individuals
Brief Title: The Association Between Sarcopenia and the Strength of Peripheral and Respiratory Muscles in Elderly Individuals
Status: Not yet recruiting | Type: Observational
Sponsor: Biruni University (Other)
Collaborators: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Associate professor, Biruni University
Other Study IDs: 202412
Record Dates: First submitted 2024-12-22; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: The Association Between Sarcopenia and the Strength of Peripheral and Respiratory Muscles in Elderly Individuals; Cardiovascular Diseases; Diabetes Mellitus; Hypertension
Keywords: Muscle strength, respiratory muscle strength, sarcopenia .; Cardiovascular diseases; Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Hypertension; Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly Individuals: The study group was composed of volunteers aged 65-80 years.
  Interventions: Other: Questionnare, hand grip and respiratory muscle strength

INTERVENTIONS:
Other: Questionnare, hand grip and respiratory muscle strength — Upper extremity strength will be assessed using the Jamar hand dynamometer to measure hand grip strength. For lower extremity muscle strength, participants will undergo the five-repetition sit-to-stand test. Respiratory muscle strength, both inspiratory and expiratory, will be measured through mouth pressure assessments. Additionally, participants will complete a questionnaire addressing components related to sarcopenia diagnosis, including questions on strength, assistance with walking, rising from a chair, climbing stairs, and incidence of falls.

SUMMARY:
Population aging is a significant global trend, with projections indicating that by 2050, 1 in 6 individuals worldwide will be over 65 years old, compared to 1 in 11 in 2019. In Turkey, the elderly population is expected to rise to 11.0% by 2025 and reach 25.6% by 2080. Sarcopenia, characterized by the progressive loss of skeletal muscle mass (SMM) and function due to aging, affects approximately 29% of older adults in community healthcare settings. It is associated with various pathophysiological processes, leading to negative health outcomes like falls and frailty.

The European Working Group on Sarcopenia in Older People (EWGSOP) established diagnostic criteria for sarcopenia based on muscle mass, strength, and physical performance in 2010, later revised in 2018 (EWGSOP2), emphasizing low muscle strength as the primary diagnostic criterion. The SARC-F questionnaire is recommended for confirming sarcopenia, with a score of ≥ 4 indicating the condition.

The concept of respiratory sarcopenia, introduced in 2021, refers to the loss of respiratory muscle mass and strength alongside general body sarcopenia, though measuring respiratory muscle mass can be complex. Respiratory muscle strength can be assessed through mouth pressure measurement, but a consensus on the methodology is still lacking.

Overall, there is insufficient research on the relationship between peripheral and respiratory muscle weakness and sarcopenia in the elderly. This study aims to explore this relationship further.

DETAILED DESCRIPTION:
Population aging is a global phenomenon characterized by a significant and rapid increase in the elderly population over recent years. According to World Population Prospects 2019 (United Nations, 2019), by 2050, 1 in 6 people in the world will be over the age of 65, up from 1 in 11 in 2019. It is estimated that the elderly population rate in our country will be 11.0% in 2025, 12.9% in 2030, 16.3% in 2040, 22.6% in 2060 and 25.6% in 2080.

Sarcopenia is a progressive and characterized loss of skeletal muscle mass (SMM) and function associated with aging. Several prospective studies have reported that skeletal muscle mass decreases by 6% per decade after middle age. In community healthcare settings, the prevalence of sarcopenia has been reported to reach up to 29% among older adults. Sarcopenia is thought to involve a variety of pathophysiological processes, including denervation, mitochondrial dysfunction, inflammatory and hormonal changes that can lead to adverse health outcomes such as falls, functional decline, frailty, weakness, and death due to a decrease in lean body mass. The European Working Group on Sarcopenia in Older People (EWGSOP) proposed three diagnostic criteria for sarcopenia based on muscle mass, muscle strength, and physical performance in 2010. The EWGSOP proposed for sarcopenia three diagnostic criteria; low muscle mass (LMM) is defined by a SMM index of less than 8.90 kg/m2, low muscle strength (LMS) by hand-grip strength below 30 kg in men and 20 kg in women, and low physical performance (LPP) by gait speeds of less than 0.8 m/s. In 2018, The European Working Group on Sarcopenia in Older People 2 (EWGSOP2) revised the diagnostic criteria and established that low muscle strength is the primary parameter for the diagnosis of sarcopenia and the most reliable measure of muscle function. In clinical practice, when a patient shows symptoms or signs of sarcopenia (i.e. falls, feeling weak, walking slowly and difficulty getting up from a chair, or weight loss or muscle wasting), the EWGSOP2 is recommended to use the SARC-F questionnaire, which consists of five items: Strength, Assistance in walking, Rising from a chair, Climbing stairs, and Falls to confirm the diagnosis. A score of the SARC-F questionnaire ≥ 4 is considered sarcopenia.

The concept of respiratory sarcopenia was first proposed in 2021 and is defined as "General body sarcopenia and low respiratory muscle mass followed by low respiratory muscle strength and/or low respiratory function." Diagnosis of respiratory sarcopenia is made by assessing respiratory muscle mass and strength. However, measuring respiratory muscle mass can often be complex, requiring advanced diagnostic equipment or techniques such as ultrasound echography and computed tomography. Assessing respiratory muscle strength is easier because it can be measured by mouth pressure measurement; however, there is no consensus yet on the exact methodology.

Studies showing the relationship between peripheral muscle and respiratory muscle weakness and sarcopenia in the elderly population are insufficient. In our study, we aim to examine the relationship between sarcopenia and peripheral and respiratory muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* 65 years to 80 years (Older ),
* Standardised Mini Mental Test score ≥ 20,
* Volunteering to participate in the study study
* Registered at the Çanakkale Municipality Golden Years Life Center.

Exclusion Criteria:

* With with a history of respiratory disease or receiving treatment for respiratory disease
* With serious orthopedic diseases that may affect the measurements
* Diagnosed with dementia
* Smokers.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The Çanakkale Municipality Golden Years Life Center.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-02-24 (Estimated)

PRIMARY OUTCOMES:
The sociodemographic data form | baseline
  Socio-demographic data of individuals (name-surname, age, gender, height, weight, smoking, occupation, education) will be collected with the demographic data collection form created by the researchers. In the clinical information section, other diseases and medications used will berecorded.
Hand grip strength | baseline
  Upper extremity strength will be measured by hand grip strenght with a Jamar hand dynamometer. Participants will be seated with the dynamometer in their dominant hand, elbows flexed at 90° and next to the body, and three consecutive measurements will be taken with a 1-minute interval between measurements. The highest value will be recorded.
The five-repetition sit-to-stand test | baseline
  Lower extremity muscle strength will be evaluated. Participants will test to cross their arms on their chest and sit down and stand up on a chair once for trial purposes. After the trial performance, they will be asked to sit down and stand up on the chair as quickly as possible without stopping, and the time will be recorded after the fifth repetition
Measurements of respiratory muscle strength | baseline
  Inspiratory and expiratory respiratory muscle strength will be evaluated by the mouth pressure measurement.
SARC-F questionnaire | baseline
  Participants will be asked the questionnaire about strength, assistance in walking, rising from a chair, climbing stairs, and falls components. Each component will be scored between 0-2. The total scores will be recorded that ranged from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Buket Akıncı, Ass.Prof, Principal Investigator — Biruni University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bahat G, Yilmaz O, Kilic C, Oren MM, Karan MA. Performance of SARC-F in Regard to Sarcopenia Definitions, Muscle Mass and Functional Measures. J Nutr Health Aging. 2018;22(8):898-903. doi: 10.1007/s12603-018-1067-8. PMID 30272090
- [Background] Bohannon RW. Five-repetition sit-to-stand test: usefulness for older patients in a home-care setting. Percept Mot Skills. 2011 Jun;112(3):803-6. doi: 10.2466/15.26.PMS.112.3.803-806. PMID 21853769
- [Background] Cho MR, Lee S, Song SK. A Review of Sarcopenia Pathophysiology, Diagnosis, Treatment and Future Direction. J Korean Med Sci. 2022 May 9;37(18):e146. doi: 10.3346/jkms.2022.37.e146. PMID 35535373
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Background] Malmstrom TK, Morley JE. SARC-F: a simple questionnaire to rapidly diagnose sarcopenia. J Am Med Dir Assoc. 2013 Aug;14(8):531-2. doi: 10.1016/j.jamda.2013.05.018. Epub 2013 Jun 25. No abstract available. PMID 23810110
- [Background] Ohara DG, Pegorari MS, Oliveira Dos Santos NL, de Fatima Ribeiro Silva C, Monteiro RL, Matos AP, Jamami M. Respiratory Muscle Strength as a Discriminator of Sarcopenia in Community-Dwelling Elderly: A Cross-Sectional Study. J Nutr Health Aging. 2018;22(8):952-958. doi: 10.1007/s12603-018-1079-4. PMID 30272099
- [Background] Sawaya Y, Hirose T, Ishizaka M, Shiba T, Sato R, Kubo A, Urano T. Patterns of Changes in Respiratory Muscle Strength over 1 Year in Non-Sarcopenia, Sarcopenia, and Severe Sarcopenia. Int J Environ Res Public Health. 2022 Dec 9;19(24):16571. doi: 10.3390/ijerph192416571. PMID 36554450
- [Background] Woo J, Leung J, Morley JE. Validating the SARC-F: a suitable community screening tool for sarcopenia? J Am Med Dir Assoc. 2014 Sep;15(9):630-4. doi: 10.1016/j.jamda.2014.04.021. Epub 2014 Jun 16. PMID 24947762